CLINICAL TRIAL: NCT06794047
Title: The Effect of Vitamin C Supplementation on Assisted Reproductive Pregnancy Outcomes in Patients With Diminished Ovarian Reserve: A Multicenter, Double-blind, Randomized Controlled Trial.
Brief Title: The Effect of VitC on IVF Outcome of DOR Patients
Acronym: DORIVF-VC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Obstetrics and Gynecology Hospital (Other); Peking University Shenzhen Hospital (Other); Tang-Du Hospital (Other); General Hospital of Ningxia Medical University (Other); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Jie Qiao, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M2024646; No2024 (Other Grant/Funding Number: National Clinical Research Center for Obstetrics and Gynecology, Peking University Third Hospital, China)
Record Dates: First submitted 2025-01-08; First posted 2025-01-27 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Diminished Ovarian Reserve; IVF Outcomes
Keywords: vitamin C; IVF outcomes; livebirth; diminished ovarian reserve
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the entire implementation of the RCT, a double-blind design was employed for both the study subjects and researchers. Group allocation concealment was applied to study subjects, clinical practitioners involved in the RCT, outcome observers and assessors, and subsequent data analysts. The pharmaceutical company assigned numbers and labels to the drugs, and when study subjects were enrolled, they were assigned the corresponding drug number. The specific group corresponding to the number remained concealed from the project researchers, participants, and study subjects, with the blind data kept by independent personnel.
  After the follow-up, independent personnel who maintained the blind data provided group information to the data analysts. The vitamin C and control groups were still represented as A and B, concealing the specific identities of the AB groups from the data analysts. After the data comparison between the two groups the unblinding of the AB groups was conducted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VitC (Experimental): The women will intake the vitamin C twice a day, 500mg per time.
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Tablets with the same material, flavor, and appearance as the intervention group.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — Vitamin C tablets, please instruct the patient to swallow with water, 500mg twice daily, morning and evening.
  Other Names: VitC; VC; Ascorbic acid
  Arms: VitC
Other: Placebo — Tablets with the same material, flavor, and appearance as the intervention group.
  Other Names: control
  Arms: Placebo

SUMMARY:
In the context of the accelerating aging population and the continuous decline in birth rates nationwide, delaying reproductive aging in women and protecting the fertility of women of childbearing age have become urgent issues and key demands that need to be addressed in the field of maternal and child health in China. The ovaries have reproductive and hormone secretion functions and are crucial throughout the female reproductive lifecycle. Women of childbearing age in China face a serious problem of diminished ovarian reserve (DOR), which can lead to infertility, failed in vitro fertilization (IVF) treatments, miscarriage, and other adverse pregnancy outcomes, severely affecting the safety of women and their offspring. For DOR patients who desire to conceive, failure to intervene and treat promptly can result in irreversible losses and impose a significant psychological burden on them. However, there are currently no clear and reliable interventions that can improve ovarian function and enhance fertility in women with DOR. Therefore, exploring new, safe, and patient-acceptable intervention strategies is urgently needed, as it may bring hope and light to women with DOR. Nutrient supplementation, especially vitamin supplementation, has received increasing attention in disease treatment due to its safety, bioavailability, and effectiveness. Previous studies have shown that vitamin C may play an important role in treating diminished ovarian reserve. However, its effects on ovarian function need to be validated in the population.

Based on the above research background, this project will conduct a randomized, placebo-controlled, double-blind, multicenter trial. The study subjects will be DOR infertility patients undergoing IVF/ICSI treatment. The intervention group will receive oral vitamin C supplementation at a dosage of 500 mg per dose, twice a day; the control group will receive a placebo with the same dosage and method for at least three months. Patients will be followed up until delivery outcomes, comparing the IVF/ICSI treatment results between the vitamin C supplementation group and the placebo group. The primary endpoint of this clinical trial is the live birth rate of the IVF/ICSI treatment cycle. Secondary endpoints include indicators of improved ovarian reserve function, ovarian aging molecular clocks, IVF-embryo culture indicators, pregnancy rates, pregnancy complications, and neonatal conditions, thereby providing new clues and theoretical basis for clinical treatment plans for DOR patients.

ELIGIBILITY:
Definition of DOR: Currently, there is no internationally unified standard for DOR. According to the latest POSEIDON criteria for diminished ovarian reserve (DOR), serum AMH <1.20 ng/mL or bilateral antral follicle count (AFC) <5 is classified as DOR.

In this study, the participants are primarily DOR patients, with the following inclusion criteria:

* Infertile women undergoing their 1st or 2nd IVF treatment
* Diagnosed with DOR: POSEIDON criteria (AMH <1.2 ng/mL or bilateral AFC <5) BMI between 18.5-28.0 kg/m²
* Signed informed consent

Exclusion Criteria：Participants meeting any of the following criteria will be excluded from the trial:

* PGT (preimplantation genetic testing) candidates
* DOR caused by ovarian surgery, cancer radiotherapy/chemotherapy
* Other ovulation disorders (e.g., PCOS, Cushing's syndrome, non-classic congenital adrenal hyperplasia, hyperprolactinemia) or endometriosis (chocolate cysts)
* Severe thyroid disorders: Hyperthyroidism, Graves' disease, Hashimoto's thyroiditis
* Acute/chronic renal insufficiency, hemodialysis, or history of severe kidney impairment
* Infectious diseases: HIV, active hepatitis, metabolic acidosis, tuberculosis, etc.
* Severe autoimmune diseases (e.g., rheumatoid arthritis, lupus, Crohn's disease)
* Cardiovascular events within the past 3 months: Coronary artery disease/myocardial infarction/clinically significant congestive heart failure；Stroke/transient ischemic attack (TIA)；Deep vein thrombosis/pulmonary embolism；Poorly controlled hypertension (SBP ≥160 mmHg or DBP ≥90 mmHg)；Diagnosed diabetes mellitus；Coronary intervention (PCI) or coronary artery bypass grafting (CABG)；
* Neurological disorders (e.g., dementia,Alzheimer's, Parkinson's) or use of related medications
* Psychiatric disorders or use of antiepileptic/antidepressant drugs
* History of cancer or radiotherapy/chemotherapy
* Allergy to vitamin C
* Current high-dose vitamin C supplementation (>500 mg/day)
* Unwillingness to take the study-provided supplements
* Alcohol abuse, smoking, or drug addiction
* Participation in other clinical trials within the past month

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 1 year after oocyte retrieval following embryo transfer
  The main outcome of this trial is the live birth resulting from a sustained pregnancy after the first embryo transfer within 6 months for patients undergoing fresh transfer cycles or frozen embryo cycles.
  Live birth rate (%) = Number of subjects with live births in each group / Total number of subjects in each group × 100%.

SECONDARY OUTCOMES:
Cumulative live birth rate | 1 year after oocyte retrieval following embryo transfer
  Live births within 1 year after oocyte retrieval following embryo transfer; calculated as: (Final number of live births / Number of randomized participants) × 100%
Singleton live birth rate | 1year after oocyte retrieval following embryo transfer
  (Number of singleton live births / Number of randomized participants) × 100%
Twin live birth rate | 1 year after oocyte retrieval following embryo transfer
  (Number of women with twin live births / Number of randomized participants) × 100%
Clinical pregnancy rate | 28-30 days after embryo transfer
  Presence of at least one gestational sac (including intrauterine and ectopic) confirmed by transvaginal ultrasound 28-30 days after embryo transfer; includes singleton pregnancy rate and twin pregnancy rate (twin and multiple pregnancy rates should be reported along with pregnancy loss rate)
Ongoing pregnancy | 12 weeks after embryo transfer.
  Presence of at least one gestational sac with fetal heartbeat confirmed by transvaginal ultrasound at 12 weeks after embryo transfer.
Time to pregnancy leading to live birth | 1 year after oocyte retrieval following embryo transfer
  or participants who achieved live birth, the time from intervention initiation to clinically confirmed pregnancy (confirmed by ultrasound 30 days after transfer). Survival analysis will be used to compare between intervention and control groups.
Number of oocytes retrieved | 3 to 12 months from enrollment
  Number of oocytes retrieved
Number of normally fertilized oocytes | Day 1 post-retrieval
  On Day 1 post-retrieval, oocytes with two pronuclei (2PN) are counted as normally fertilized.
Total fertilization failure | Day 1 post-retrieval
  No oocytes in the current treatment cycle show 2PN after fertilization or injection.
Number of usable embryos | On Day 3 post-retrieval
  On Day 3 post-retrieval, embryos with ≥4 cells and ≤30% fragmentation are considered usable.
Number of high-quality embryos | On Day 3 post-retrieval
  On Day 3 post-retrieval, 2PN-derived embryos with ≥6 cells and ≤10% fragmentation are classified as high-quality.
Number of implanted embryos | 28-30 days after embryo transfer.
  The number of gestational sacs (including intrauterine and ectopic) detected by transvaginal ultrasound 28-30 days after embryo transfer.
Ectopic pregnancy | 1 year after oocyte retrieval following embryo transfer
  A pregnancy occurring outside the uterine cavity, diagnosed by ultrasound, surgical visualization, or histopathology.
Miscarriage | 1 year after oocyte retrieval following embryo transfer
  Spontaneous loss of an intrauterine pregnancy before 20 weeks of gestation. This should occur after ultrasound confirmation of a viable pregnancy.
Stillbirth | 1 year after oocyte retrieval following embryo transfer
  Fetal death occurring after 20 weeks of gestation, before complete expulsion or extraction. Death is determined by the absence of breathing or other signs of life (e.g., heartbeat, umbilical cord pulsation, or definite voluntary movement) after delivery.
Termination of pregnancy | 1 year after oocyte retrieval following embryo transfer
  Medical, surgical, or other artificial termination of an intrauterine pregnancy (including fetal reduction procedures).
Moderate or severe ovarian hyperstimulation syndrome (OHSS) | 1 year after oocyte retrieval following embryo transfer
  OHSS is primarily characterized by cystic enlargement of the ovaries, increased vascular permeability, third-space fluid accumulation (resulting in ascites and pleural effusion), and localized or generalized edema.)
Pregnancy complications | 1 year after oocyte retrieval following embryo transfer
  Including gestational diabetes mellitus, hypertensive disorders of pregnancy, antepartum hemorrhage, etc.
Gestational age | 1 year after oocyte retrieval following embryo transfer
  The number of weeks from fertilization to delivery, plus 14 days.
Preterm birth | 1 year after oocyte retrieval following embryo transfer
  Birth occurring before 37 weeks of gestation (i.e., fewer than 259 days of pregnancy).
Birth weight | 1 year after oocyte retrieval following embryo transfer
  The weight of the newborn at birth. Abnormal birth weight includes: Low birth weight (LBW): <2,500 g Very low birth weight (VLBW): <1,500 g High birth weight (macrosomia): >4,000 g Very high birth weight: >4,500 g
Large for gestational age (LGA) | 1 year after oocyte retrieval following embryo transfer
  Newborns with birth weight above the 90th percentile for their gestational age and sex.
Small for gestational age (SGA) | 1 year after oocyte retrieval following embryo transfer
  Newborns with birth weight below the 10th percentile for their gestational age and sex.
Neonatal death | 1 year after oocyte retrieval following embryo transfer
  Death of a live-born infant within 28 days after birth. This can be further categorized as:
  Early neonatal death: Death occurring within the first 7 days of life. Late neonatal death: Death occurring between 8 and 28 days of life.
Birth defect | 1 year after oocyte retrieval following embryo transfer
  Structural, functional, or genetic abnormalities occurring during pregnancy, which may be identified prenatally, at birth, or postnatally, and may be life-threatening or fatal. Major congenital anomalies should be reported as infants with at least one major congenital anomaly detected. If a major birth defect is identified in a multiple pregnancy, it should be explicitly reported.
Possible Vitamin C Side Effects-Abdominal Pain and Diarrhea: | 1 year
  A single high dose (5-10 g) of vitamin C may cause transient osmotic diarrhea and/or abdominal bloating. However, the human body has a high tolerance, and even such high doses are generally safe. Typically, these symptoms gradually improve or disappear after continued use.
Possible Vitamin C side effect--Hyperuricemia | 1 year
  Hyperuricemia: Vitamin C can be partially metabolized into oxalate and dose-dependently increase oxalate levels in urine. High doses of vitamin C may temporarily increase uric acid excretion, while high-dose intravenous administration may stimulate polyuria. Therefore, the daily recommended dose of vitamin C should not exceed 1 gram. Urine routine tests will be conducted during follow-up.
Possible Vitamin C side effect--Kidney stones | 1 year
  Some studies have found that high-dose oral vitamin C significantly increases the risk of kidney stone formation in men by 41%. Additionally, long-term high concentrations of oxalate in urine may contribute to stone formation. Thus, high-dose vitamin C supplementation in at-risk populations may lead to urinary tract stones, as self-reported by participants.
Possible Vitamin C side effect--Hemolysis | 1 year
  Intravenous or high-dose oral vitamin C may induce hemolysis in patients with glucose-6-phosphate dehydrogenase (G6PD) deficiency and worsen hemolysis in those with paroxysmal nocturnal hemoglobinuria. If such symptoms occur, vitamin C should be discontinued immediately, medical attention sought, and researchers contacted.
Vitamin C level after supplementation | 3 months to 1 year

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Obstetrics and Gynecology Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Peking university third hospital, Beijing, Beijing Municipality
  - The second hospital of Hebei Medical University, Shijiazhuang, Hebei
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Tang Du Hospital, Xi’an, Shanxi
  - Peking University Shenzhen Hospital, Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: No
We have decided not to share the IPD from this study due to concerns about participant privacy and confidentiality. Despite efforts to de-identify the data, there remains a risk of re-identification, which could compromise the privacy of the participants involved. Additionally, there are legal and ethical considerations that restrict the sharing of sensitive health information without explicit consent from the participants. Furthermore, the resources required to prepare and manage the data for external sharing are currently beyond our capacity. Therefore, to ensure the protection of our participants and comply with ethical standards, we have opted not to share the IPD at this time.